CLINICAL TRIAL: NCT01330706
Title: Efficacy of Intraoperative Surgical Scrubbing in Reducing Bacterial Load After Nail Removal Surgery
Acronym: ribebeva
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Ricardo Becerro de Bengoa Vallejo, Universidad Complutense de Madrid
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UCM 2011
Record Dates: First submitted 2011-04-01; First posted 2011-04-07 (Estimated); Last update posted 2011-04-07 (Estimated); Status verified 2009-02

CONDITIONS: Skin Diseases; Nail Diseases; Nails, Ingrown
Keywords: Skin Diseases [C17.800]; Nail Diseases [C17.800.529]; Nails, Ingrown [C17.800.529.406]
MeSH Terms: conditions — Skin Diseases; Nail Diseases; Nails, Ingrown | interventions — polihexanide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sterile Saline solution (Experimental): The investigators compared intraoperative antiseptic irrigation using 0.9% saline solution and 0.1% polihexanide.
  Interventions: Drug: Polihexanide

INTERVENTIONS:
Drug: Polihexanide — The investigators compared intraoperative antiseptic irrigation using 0.9% saline solution and 0.1% polihexanide.

SUMMARY:
The investigators conducted a controlled, prospective randomized study to examine the antiseptic efficacy of intraoperative irrigation methods during nail avulsion surgery.

DETAILED DESCRIPTION:
The investigators conducted a controlled, prospective randomized study to examine the antiseptic efficacy of intraoperative scrubbing methods during nail avulsion surgery. The investigators compared intraoperative antiseptic scrubbing using 0.9% saline solution and 0.1% polihexanide. Swab samples were taken from each patient at 5 distinct stages throughout the surgical procedure, and bacterial culture analysis was performed (positive culture rate, total inocula count, reduction of bacterial load, and identification of specific microorganisms).

ELIGIBILITY:
Inclusion Criteria:

* Older than 18
* Onychocryptosis

Exclusion Criteria:

* infection
* a history of tinea pedis
* onychomycosis
* paronychia
* nail trauma or subungual hematoma
* nail deformities and disorders
* peripheral vascular disease or diabetes
* cardiac disease
* a history of rheumatic fever
* recent antibiotic use or current antimicrobial therapy
* a history of steroid use and
* recent nail polish use

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-02; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
bacterial count (CFU/cm2) | Participants will be followed until the surgery to heal completely,an expected average of 7 weeks
  The percentage of inoculum reduction at the irrigation step was calculated as follows: percentage of inoculum reduction = 100 e (1003 Ii)/Is, where Ii is the bacterial count (CFU/cm2) at the irrigation step and Is is the inoculum (CFU/cm2) at the surgery step.
  Bacteria were identified using standard laboratory methods. The limit of detection in the nailfold test was 1.33 CFU/cm2.

CONTACTS AND LOCATIONS:
Overall Officials: Ricado Becerro de Bengoa Vallejo, PhD, Principal Investigator — Universidad Complutense de Madrid
Locations (1):
- Universidad Complutense de Madrid, Madrid, Madrid, Spain

REFERENCES:
- [Background] Becerro de Bengoa Vallejo R, Losa Iglesias ME, Cervera LA, Fernandez DS, Prieto JP. Efficacy of intraoperative surgical irrigation with polihexanide and nitrofurazone in reducing bacterial load after nail removal surgery. J Am Acad Dermatol. 2011 Feb;64(2):328-35. doi: 10.1016/j.jaad.2010.01.011. Epub 2010 Nov 26. PMID 21112671
- See also: University Complutense de Madrid — http://www.ucm.es